CLINICAL TRIAL: NCT04610268
Title: Mechanism Study of tDCS on Human Electrophysiological Network Via SEEG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Qiushi Academy for Advanced Studies, Zhejiang University (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-145
Record Dates: First submitted 2019-07-19; First posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-09

CONDITIONS: Depression
Keywords: Transcranial direct current stimulation (tDCS); Stereotactic electroencephalography (sEEG); Focal refractory epilepsy
MeSH Terms: conditions — Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tDCS group (Experimental): The anode of tDCS is placed on the occipital lobe and the cathode on the frontal lobe, or the anode of tDCS is placed on the left temporal lobe and the cathode on the right temporal lobe.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Depending on the location of sEEG electrode implanted in the patient's head, the tDCS electrode (5 cm×7 cm each) was placed on occipital-frontal lobe or bilateral temporal lobe. Current intensity: 2 mA and 4 mA, Stimulus time: 3 min (each stimulus session).

SUMMARY:
Transcranial direct current stimulation(tDCS) is a non-invasive Neuromodulation method.The weak direct current produced by tDCS can be transmitted through the skull and induce biphase, polarization-related changes in the cortex. Related clinical studies have found that tDCS has a corresponding therapeutic effect on neurological and psychiatric diseases such as stroke rehabilitation, depression, pain, epilepsy, etc.

Stereotactic electroencephalography(sEEG) implants a set of deep electrodes into the brain that use stereotactic localization to detect electrical activity, locate epileptic foci and functional areas, and detect changes in electrical fields caused by tDCS in the deep brain. This direct measurement technology will provide validation and optimization for the electric field simulation method based on finite element analysis (FEM), also complement the latest indirect current density intensity measurement technology based on MRI phase measurement, providing support for the targeting and personalized treatment of tDCS technology.

In order to achieve this goal and study the mechanism and function of tDCS better , this project aims to realize the clinical use of sEEG to measure the electric field information generated by tDCS in the human brain in vivo.

DETAILED DESCRIPTION:
The core research objective of this project is to measure the distribution of electric field generated by tDCS in the human brain in vivo using clinical sEEG technology, and to study the influence of different tDCS stimulation parameters on the distribution of intracranial electric field intensity, so as to provide scientific basis for evaluating the effectiveness of tDCS, optimizing the stimulation parameters of tDCS, and realizing the individuation of tDCS. The project involves many scientific issues and key technologies such as "stimulus recording platform construction -- clinical trial design -- comparative research method". The main research contents are as follows.

1. Transcranial electrical stimulation and intracranial space electric field measurement system based on sEEG and tDCS.

   Multi-channel transcranial direct current stimulation technology is studied to realize the integration of parameters setting, constant current output, overcurrent protection, electrode connection status detection and other modules. Based on sEEG intracranial electric field measurement system, weak electric field measurement with spatial positioning information can be realized accurately. The integrated control system of transcranial electric stimulation and intracranial space electric field recording was studied to realize the linkage control of multi-channel tDCS and space electric field recording and data processing and analysis.
2. Clinical implementation protocol design of tDCS combined with sEEG.

   To study the implementation protocol of tDCS combined sEEG applicable to clinical practice, and to develop inclusion and exclusion criteria for clinical volunteers, based on MRI data and actual disease conditions of volunteers, individual differentiation planning of sEEG implantation and stimulation parameters and stimulation sites of combined tDCS; Intraoperative sEEG-based intracranial spatial electric field measurement protocols were studied, including implementation procedures for tDCS stimulation and sEEG recording, individualized experimental paradigm design, practical procedures and data recording.
3. Individual head model electric field simulation analysis method.

An electric field distribution simulation model based on individual head model was established to realize the finite element simulation calculation of spatial electric field distribution under different individual head model structure, different electrical properties of tissues, different tDCS stimulation combinations and stimulation parameters. According to the electric field data recorded by sEEG and MRI data, the actual electric field distribution model of individual head model was established. The spatial electric field distribution characteristics of tDCS acting on different intracranial depths and distances were analyzed under different external stimulation parameters, and compared with the simulation model. The existing simulation model is optimized based on the measured data.

ELIGIBILITY:
Inclusion Criteria:

* SEEG is required for preoperative evaluation in patients with focal refractory epilepsy, consent and sign the informed consent for treatment.

Exclusion Criteria:

* (1) history of major depression or mental disorder and medication history causing symptoms of mental disorder,
* (2) patients with severe cognitive impairment (MMSE score<17),
* (3) craniocerebral surgery history,
* (4) severe head skin disease (including but not limited to purpura, blisters, rash, eczema) or open head injury/laceration,
* (5) existing known risk factors of tDCS: A. use of implanted electronic devices (such as pacemakers) or metal implants (such as stents), B. a history of injury to unfixed metal in any part of the body (including metal objects in the eye), C. pregnant woman;D. cancer patients, patients in critical condition or patients with important organ failure, E. severe allergy to the electrode patch, local skin injury or inflammation, and hyperalgesia in the stimulation area, F. scalp injury that may cause poor application of tDCS.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Voltage difference | intraoperative
  Voltage difference between stimulation electrodes.
Stimulus current | intraoperative
  Stimulus current between stimulation electrodes.
sEEG voltage | intraoperative
  Respectively, 2 to 4 sEEG electrodes with distance of more than 2 cm were selected along the sagittal plane direction and coronal plane direction, and the voltage of each channel on the electrode was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Hongjie Jiang, Dr., Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- SAHZhejiangU, Hangzhou, Zhejiang, China